CLINICAL TRIAL: NCT00410358
Title: A Phase I Dose Escalation Study of LBQ707 (Gimatecan) Administered Orally 5 Consecutive Days to Japanese Patients With Advanced Solid Tumor.
Brief Title: A Dose Escalation of Gimatecan Administered Orally to Japanese Patients With Advanced Solid Tumor.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBQ707A1101
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2012-10

CONDITIONS: Advanced Solid Tumors
Keywords: Gimatecan; topoisomerase I inhibitor; advanced solid tumors
MeSH Terms: interventions — ST 1481

ARMS (1):
- LBQ707 (Experimental)
  Interventions: Drug: Gimatecan

INTERVENTIONS:
Drug: Gimatecan
  Other Names: LBQ707

SUMMARY:
This study assesses the tolerability, safety, efficacy and pharmacokinetics of gimatecan in Japanese patients. Gimatecan is administered orally for five consecutive days, every 28 days, to adult patients with advanced solid tumors who have progressed despite standard therapy or for whom standard systemic therapy does not exist.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological or cytological confirmed advanced solid tumors, which have progressed despite standard therapy or for whom no standard therapy exists.
* Life expectancy of at least 3 months
* Adequate hematological parameters
* No major impairment of renal and hepatic function

Exclusion Criteria:

* Gastrointestinal dysfunction, such as gastrectomy and malabsorption syndrome that could alter absorption.
* Patients who have received any investigational compound within the past 28 days.
* Patients with other antineoplastic therapy within the last 28 days.
* Patients known to be HIV or hepatitis virus positive, or patients with the presence of active or suspected acute or chronic uncontrolled infection
* Patients with a history of allergies to the camptothecin family drug.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-06; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Estimated Maximum Tolerated Dose of gimatecan | 1.8 years

SECONDARY OUTCOMES:
Safety assessed by adverse events | 1.8 years
Characterization of the pharmacokinetic profile of gimatecan | 1.8 years
Anti-tumor activity assessed by RECIST | 1.8 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Chiba Prefecture, Japan

REFERENCES:
- See also: Results for CLBQ707A1101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3945